CLINICAL TRIAL: NCT03715738
Title: MEasurement by a Numerical Approach of BREAst Volume MENABREA
Brief Title: MEasurement by a Numerical Approach of BREAst Volume
Acronym: MENABREA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-A02018-47
Record Dates: First submitted 2018-08-30; First posted 2018-10-23 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Breast Asymmetry, 3D
MeSH Terms: conditions — Anisomastia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- arm 1 : Creaform3D + MyotonPRO (Experimental): A clinical questionnaire is completed by the investigator (chest circumference, thorax turn, breast "measurements").
  The breast density is assessed by the surgeon and scored from 1 to 5 (Likert scale) and then by the MyotonPRO The volumetric measurement of the breast is performed using the 3D digital camera. The patient is bent forward with hands resting on a chair during 30 seconds to 1 minute. The 3D digital camera rotates around the breast to capture the volume of the breast.
  Intraoperatively, the weight of tissues removed is weighed (in grams), recorded in the observation notebook.
  In post-operative (4 months), the possible long-term complications related to the intervention (mainly the dissatisfaction of the patient as for the aesthetic result) are collected then a new acquisition of the mammary volume is carried out with the digital camera 3D.
  Once this measurement is completed, participation in the study is complete
  Interventions: Other: arm 1 : Creaform3D + MyotonPRO

INTERVENTIONS:
Other: arm 1 : Creaform3D + MyotonPRO — After inclusion,are carried out:
  * estimation of the volume of the breast to be reduced with the 3D digital camera
  * measurement of breast density by Likert scale and MyotonPRO
  The volumetric measurement of the breast is performed using the 3D digital camera. The patient is bent forward with hands resting on a chair to be as still as possible over a period of 30 seconds to 1 minute. The 3D digital camera rotates around the breast to capture the volume of the breast.
  In peroperative, the weight of tissues removed is weighed (in grams). The removed weight is recorded in the observation notebook.
  In postoperative (4 months), the possible long-term complications related to the intervention (mainly the dissatisfaction of the patient as for the aesthetic result) are collected then a new acquisition of the mammary volume is carried out with the digital camera 3D.
  Once this measurement is completed, participation in the study is complete.

SUMMARY:
Breast asymmetry is a rare in plastic surgery. In majority of cases, it is idiopathic.

In cases that are poorly tolerated physically (vertebral imbalance, posture disorders) or psychologically, the decision to perform breast symmetrization surgery can be made. It is recommended to do this surgery after a slimming treatment if the woman is overweight or after pregnancy that causes a change in the structure and volume of the chest. In fact, the weight variations deteriorate the long-term result.

However, this surgical management remains difficult. In fact, the volume to be removed (unilateral breast reduction) to be symmetrized is a function of the volume of the contralateral breast and the preoperative drawings are made while standing. Currently, the evaluation of the volume to be removed remains subjective and is based on the experience of the surgeon. In addition, intraoperatively, this evaluation is also subjective because the patient is lying down which changes the position of the anatomical landmarks: the optimization of the symmetrization is only possible by the eye and the touch.

No measuring device is currently used to assess the difference in volume between the 2 breasts and guide the surgeon in the volume (or weight) to remove. It is therefore sometimes necessary to perform a second intervention in case of residual postoperative asymmetry.

Primary objective :

To study the association between the weight of tissues removed during the intervention and the variation of the breast volume (pre / postoperative) measured by the Créaform® GOPRO 3D digital camera adjusted on the density of the gland measured by electronic palpation (MyotonPRO).

Second objective : To study the association between the weight of tissues removed during the procedure and the variation of the breast volume (pre / postoperative) measured by the Créaform® GOPRO 3D digital camera adjusted on the density of the gland estimated by manual palpation (Likert scale from 1 to 5).

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for uni / bilateral breast reduction as part of an indication of surgical management.
* Major patients.
* Patients affiliated or beneficiaries of a social security scheme
* Patients who have signed prior informed consent.

Exclusion Criteria:

* Protected patients (pregnant, parturient and lactating women, persons deprived of their liberty by an administrative or judicial decision, persons undergoing psychiatric care under duress, minors, adults over the age of 18) legal protection measure or unable to express their consent).
* Patients unfit to understand the objectives or instructions of the study.
* Patients in an exclusion period relative to another interventional study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
association between weight and volume adjusted to the density of the gland measured by electronic palpation | one year
  To study the association between the weight of tissues removed during the intervention and the variation of the breast volume (pre / postoperative) measured by the Créaform® GOPRO 3D digital camera adjusted on the density of the gland measured by electronic palpation (MyotonPRO).
  Primary judgment criterion:
  Coefficient associated with volume variation in the linear regression model (model 1) explaining weight by volume variation and density measured by electronic palpation.

SECONDARY OUTCOMES:
association between weight and volume adjusted to the density of the gland estimated by manual palpation | one year
  To study the association between the weight of tissues removed during the procedure and the variation of the breast volume (pre / postoperative) measured by the Créaform® GOPRO 3D digital camera adjusted on the density of the gland estimated by manual palpation (Likert scale from 1 to 5).
  Secondary judgment criterion 1:
  Coefficient associated with volume variation in the linear regression model (Model 2) explaining weight by volume variation and estimated density by manual palpation.
comparison of models 1 and 2 | one year
  Comparison of models 1 and 2 (estimated density by manual palpation or measured by electronic method), to see if one model is better than the other.
  Secondary judgment criterion 2:
  Akaike Criterion

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, Maine Et Loire, France

IPD SHARING:
Plan to Share IPD: No